CLINICAL TRIAL: NCT04035265
Title: Application of MRI for Inflammatory Musculoskeletal Involvement in Systemic Lupus Erithematosus (SLE)
Brief Title: Application of MRI for Musculoskeletal Involvement in SLE
Acronym: RMNLES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Patricia Corzo, M.D. Rheumatologist consultant, Hospital del Mar
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RMNLES
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Hand Rheumatism; Systemic Lupus Erythematosus Arthritis
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: 1. Lupus with synovitis
  2. Lupus with joint pain
  3. Lupus without synovitis/joint pain
  4. Healthy subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- pain+ / synovitis + (Active Comparator): SLE patients with inflammatory pain and synovitis determined by the practitioner during physical examination of radius and ulna carpal joint and/or carpus and/or metacarpophalangeal joint and/or IP. Defining synovitis as pain and inflammation and/or deformity (present or existing over the past year) included in the clinical history
  Interventions: Procedure: Blood test
- pain + / synovitis - (Active Comparator): SLE patients with inflammatory pain without determined synovitis. Current (or over the past year) pain in radius and ulna carpal joint and/or carpus and/or metacarpophalangeal joint and/or IP, with no synovitis
  Interventions: Procedure: Blood test
- pain - / synovitis - (Active Comparator): SLE patients without inflammatory pain with normal physical examination currently or over the past year
  Interventions: Procedure: Blood test
- healthy (Placebo Comparator): control patients (healthy participants: no pain, no SLE, no family affected by systemic inflammatory disease, a blood test with no elevation APR or autoimmunity +)
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — Carpus and fingers of non-dominating hand MRI with gadolinium contrast
  Other Names: hand MRI

SUMMARY:
Articular involvement can reach up to 95% within the chronic multisystemic manifestations of SLE (1). Originally, a non-erosive pattern of articular inflammation was described, but the emergence of more sensitive imaging techniques, such as MRI (2, 3), show synovitis, erosions (hand: 47-48%, carpus 82-84% in SLE; and hand: 18%, carpus 97% in healthy individuals), bone oedema (hand: 4-5%, carpus 13-16% in SLE; and 0% in healthy individuals) and tenosynovitis (hand 47%, carpus 79%; not evaluated in healthy individuals) in patients with SLE (4, 5). Nowadays, a specific validated pattern of articular involvement associated with this disease does not yet exist, although it has begun to be studied. This research tries to evaluate the presence, frequency and distribution of inflammatory articular manifestations in SLE (erosions, bone oedema, synovitis or tenosynovitis) using MRI (6), with the objective of trying to establish a specific pattern for this disease, if it exists, that can shorten the diagnostic process. Moreover, it tries to characterise, if they exist, clinical differences between various patient groups according to their articular involvement.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

* Nowadays no valid classification system for SLE-related arthritis/tenosynovitis exists.
* Data are not sufficient to establish an SLE-specific pattern of inflammatory involvement, similar to the pattern known for other inflammatory diseases such as rheumatoid arthritis (RA).
* Erosive arthritis associated with SLE has been typically related to patients that meet the criteria both for SLE and RA - syndrome known as Rhupus; but only a few data exist that classify erosive involvement of articular inflammation of pure SLE.
* No research exists that links the articular inflammatory pathology associated with SLE with its effect on quality of life (degree of fatigue and HAQ) or with the rest of manifestations and comorbidities associated with SLE.
* Being able to predict the development of SLE-related arthritis/tenosynovitis would be very useful when it comes to establishing the clinical management, treatment and prognosis of patients with SLE.

OBJECTIVES

* GENERAL:

  - To describe the kind of inflammatory articular involvement (synovitis/erosions/bone oedema/tenosynovitis) (6,7) and its frequency in patients affected by pure SLE (excluding Rhupus, mixed connective tissue disease, overlap syndromes).
* SPECIFIC:

  * To propose, if possible, an SLE-specific typical pattern of articular involvement.
  * To establish clinical and serological differences (extra-articular manifestations, autoimmunity, treatment received, comorbidities and quality of life) according to the type of inflammatory articular involvement and in comparison to healthy individuals.
  * To evaluate the possible link between SLEDAI/SLICC scores and the involvement using MRI.

HYPOTHESIS

* Patients with SLE have a specific inflammatory articular disease.
* A SLE-specific pattern of articular involvement exists.
* There are clinical and serological differences depending on the different patterns of articular involvement in SLE.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by SLE (1982 revised criteria) with scheduled visits to the SLE specialized medical office at Hospital del Mar:

  * (pain+ / synovitis +): SLE patients with inflammatory pain and synovitis determined by the practitioner during physical examination of radius and ulna carpal joint and/or carpus and/or metacarpophalangeal joint and/or IP . Defining synovitis as pain and inflammation and/or deformity (present or existing over the past year) included in the clinical history
  * (pain + / synovitis -) SLE patients with inflammatory pain without determined synovitis . Current (or over the past year) pain in radius and ulna carpal joint and/or carpus and/or metacarpophalangeal joint and/or IP, with no synovitis
* (pain - / synovitis -) SLE patients without inflammatory pain with normal physical examination currently or over the past year
* Control patients, without SLE nor immediate relatives affected by systemic inflammatory diseases, who lack articular pain and have blood test with no elevation APR or autoimmunity +)

Exclusion Criteria:

* Jaccoud's arthropaty
* RF + and/or ACPA +
* Incomplete SLE, MCTD, overlap syndromes
* Hand surgery
* Current neoplasia
* Non-rheumatoid systemic autoimmune diseases
* Contraindication for MRI

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
MRI inflamatory changes | 1 to 2 months after clinical assesment
  synovitis, erosions, bone oedema, tenosynovitis
SLE activity scale | at clinical assesment
  Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Measures last 10 days disease activity (rating (Y/N) 24 items related to specific manifestations on 9 organs) From 0 (best) to 105 (worst)
SLE treatments used | at clinical assesment
  Number (n and %) of participants using any approved treatments for SLE used since diagnosis
Fatigue | 2 weeks before the performance of MRI
  Fatigue Severity Scale (FSS-9) Results from 9 (best) to 63 (worst): rating 9 items ranging from 1(best) to 7 (worst)
Quality of life scale | 2 weeks before the performance of MRI
  modified health assessment questionnaire (MHAQ): Results from 0 (best) to 3 (worst): rating 9 items from 0 (best) to 3 (worst) (results given divided by 8)
SLE damage scale | at clinical assesment
  Systemic Lupus International Collaborating Clinics (SLICC) damage index:
  Irreversible damage rated by: 42 items related to 12 organs: 0 (absent-best)/1 (present-worst), some of them can count 2 or 3 (worst) if recidivant.
  From 0 (best) to 46 (worst)

SECONDARY OUTCOMES:
Serological markers of disease activity: antinuclear antibodies (ANA) | 6 months prior to 6 months after assesment
  ANA (dilution): given by titters (average titters comapred between groups)
Systemic SLE manifestations | at clinical assesment
  presence of renal, lung, skin, neurological, haematological manifestations since diagnostic (Yes/No)
Hand pain visual analogue scale (VAS) | at clinical assesment
  VAS 0 (none) to 10 (maximum)
Serological markers of disease activity: Anti-double stranded DNA antibody (DNAds) | 6 months prior to 6 months after assesment (the closest to MRI)
  Titters DNAds (UI/ml)
Serological markers of disease activity: Anti-Smith antibodies (Sm) | 6 months prior to 6 months after assesment (the closest to MRI)
  Presence of Sm (Yes/No)
Serological markers of disease activity: complement 3 (C3) | 6 months prior to 6 months after assesment (the closest to MRI)
  titters C3 (mg/dL)
Serological markers of disease activity: complement 4 (C4) | 6 months prior to 6 months after assesment (the closest to MRI)
  titters C4 (mg/dl)
Serological markers of disease activity: erythrocyte sedimentation rate (ESR) | 6 months prior to 6 months after assesment (the closest to MRI)
  ESR (mm/h)
Serological markers of disease activity: C reactive protein (CRP) | 6 months prior to 6 months after assesment (the closest to MRI)
  CRP (mg/dl)
Serological markers of disease activity:white cell blood count (WCBC) | 6 months prior to 6 months after assesment (the closest to MRI)
  WCBC: cellsx10E9/L

CONTACTS AND LOCATIONS:
Overall Officials: PAtricia corzo, MD, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will be used for PhD investigations. IPD will not be shared with other researchers

REFERENCES:
- [Background] Ball EM, Bell AL. Lupus arthritis--do we have a clinically useful classification? Rheumatology (Oxford). 2012 May;51(5):771-9. doi: 10.1093/rheumatology/ker381. Epub 2011 Dec 15. PMID 22179731
- [Background] Mosca M, Tani C, Carli L, Vagnani S, Possemato N, Delle Sedie A, Cagnoni M, D'Aniello D, Riente L, Caramella D, Bombardieri S. The role of imaging in the evaluation of joint involvement in 102 consecutive patients with systemic lupus erythematosus. Autoimmun Rev. 2015 Jan;14(1):10-5. doi: 10.1016/j.autrev.2014.08.007. Epub 2014 Aug 23. PMID 25183245
- [Background] Tani C, D'Aniello D, Possemato N, Delle Sedie A, Caramella D, Bombardieri S, Mosca M. MRI pattern of arthritis in systemic lupus erythematosus: a comparative study with rheumatoid arthritis and healthy subjects. Skeletal Radiol. 2015 Feb;44(2):261-6. doi: 10.1007/s00256-014-2033-0. Epub 2014 Oct 24. PMID 25341505
- [Background] Boutry N, Hachulla E, Flipo RM, Cortet B, Cotten A. MR imaging findings in hands in early rheumatoid arthritis: comparison with those in systemic lupus erythematosus and primary Sjogren syndrome. Radiology. 2005 Aug;236(2):593-600. doi: 10.1148/radiol.2361040844. Epub 2005 Jun 21. PMID 15972342
- [Background] Ostergaard M, Peterfy C, Conaghan P, McQueen F, Bird P, Ejbjerg B, Shnier R, O'Connor P, Klarlund M, Emery P, Genant H, Lassere M, Edmonds J. OMERACT Rheumatoid Arthritis Magnetic Resonance Imaging Studies. Core set of MRI acquisitions, joint pathology definitions, and the OMERACT RA-MRI scoring system. J Rheumatol. 2003 Jun;30(6):1385-6. PMID 12784422
- [Background] Haavardsholm EA, Ostergaard M, Ejbjerg BJ, Kvan NP, Kvien TK. Introduction of a novel magnetic resonance imaging tenosynovitis score for rheumatoid arthritis: reliability in a multireader longitudinal study. Ann Rheum Dis. 2007 Sep;66(9):1216-20. doi: 10.1136/ard.2006.068361. Epub 2007 Mar 28. PMID 17392347